CLINICAL TRIAL: NCT01948908
Title: Optimal Volumes of Administration for Intranasal Midazolam in Children
Brief Title: Volumes of Administration for Intranasal Midazolam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAL7510
Record Dates: First submitted 2013-06-29; First posted 2013-09-24 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Children Requiring Sedation to Facilitate Laceration Repair
Keywords: Sedation; Laceration repair; Children; Intranasal; Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200 mcL VOA (Experimental): Intranasal midazolam administered in 200 mcL VOA
  Interventions: Drug: Intranasal midazolam
- 500 mcL VOA (Experimental): Intranasal midazolam administered in 500 mcL VOA.
  Interventions: Drug: Intranasal midazolam
- 1000 mcL VOA (Experimental): Intranasal midazolam administered in 1000 mcL VOA.
  Interventions: Drug: Intranasal midazolam

INTERVENTIONS:
Drug: Intranasal midazolam — Intranasal midazolam, 0.5 mg/kg, maximum dose 10 mg, administered using mucosal atomization device (MAD).
  Other Names: No other name

SUMMARY:
The purpose of this study is to determine exactly how much drug volume should be administered into each nare, so that the drug absorption can be maximized and the amount that runs out of the nose, or is swallowed, is minimized, thereby optimizing the effectiveness of any drug given intranasally. The investigators will determine this ideal "volume of administration" by studying intranasal midazolam in children who require sedation to facilitate laceration repairs. The investigators will evaluate both clinical outcomes as well as pharmacokinetic outcomes associated with each volume of administration. We will block randomize children to receive intranasal midazolam in maximum aliquots of one of the three following VOA: 200 microliters (mcL), 500 mcL, or 1000 mcL.

DETAILED DESCRIPTION:
The intranasal route is an effective means of administering sedative medications for children. However, sometimes the child has to receive a certain dose that requires a very large volume to be administered into the nose, because of the types of concentrations of drugs that are available. Most drugs are not concentrated enough so that small volumes can be consistently given, so as a result, sometimes a very large amount of medication is administered intranasally. When the amount is too large, most of the medication either runs back out the nose, or down the back of the nose and throat and is swallowed, instead of being absorbed in the nasal cavity, where it can be quickly absorbed and produce optimal effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 1 to 7 years of age, inclusive.
* Require intranasal midazolam for minimal sedation to facilitate laceration repair.

Exclusion Criteria:

* Weight less than 10 kg.
* Known allergy to midazolam.
* Presence of intranasal obstruction (e.g. mucous or blood) that cannot be readily cleared
* Inability to speak English or Spanish
* Developmental delay, psychiatric illness, neurologic impairment, or altered mental status; or illnesses associated with chronic pain (e.g. sickle cell disease, inﬂammatory bowel disease).
* Foster children or wards.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States

REFERENCES:
- [Result] Tsze DS, Ieni M, Fenster DB, Babineau J, Kriger J, Levin B, Dayan PS. Optimal Volume of Administration of Intranasal Midazolam in Children: A Randomized Clinical Trial. Ann Emerg Med. 2017 May;69(5):600-609. doi: 10.1016/j.annemergmed.2016.08.450. Epub 2016 Nov 4. PMID 27823876

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200 mcL VOA | 500 mcL VOA | 1000 mcL VOA
Started | 33 | 33 | 33
Completed | 32 | 33 | 31
Not Completed | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mcL VOA | 500 mcL VOA | 1000 mcL VOA | Total
Number analyzed (Participants) | 32 | 33 | 31 | 96
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3 [2.4 to 5.6] | 2.7 [2.1 to 3.5] | 2.7 [1.9 to 3.9] | 2.9 [2 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 12 | 32
  Male | 20 | 25 | 19 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 22 | 25 | 25 | 72
  Non-Hispanic, White | 6 | 5 | 5 | 16
  Non-Hispanic, Black | 3 | 2 | 1 | 6
  Non-Hispanic, Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Time (Minutes) After Administration of Intranasal Midazolam Until Patient Achieves Minimal Sedation
Description: This outcome is designed to examine time to onset of minimal sedation, defined as a University of Michigan Sedation Score (UMSS) of 1.
Time Frame: 20 minutes
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 200 mcL VOA | 500 mcL VOA | 1000 mcL VOA
Number analyzed (Participants) | 32 | 33 | 31
minutes | 4.7 [3.8 to 5.4] | 4.3 [3.9 to 4.9] | 5.2 [4.6 to 7]

2. Secondary Outcome: Observational Scale of Behavioral Distress - Revised
Description: The Observational Scale of Behavioral Distress - revised (OSBD-r) is an eight-factor, weighted observational scale used to measure distress associated with medical procedures in children 1 to 20 years of age. The total OSBD-r score is the sum of the OSBD-r scores for predetermined clinically relevant phases of the procedure, with each phase assigned a score from 0 to 23.5 (0=no distress, 23.5=maximum distress), based on the frequency and types of behaviors observed during a pre-determined number of 15-second intervals during each phase.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: units
Arm/Group | 200 mcL VOA | 500 mcL VOA | 1000 mcL VOA
Number analyzed (Participants) | 32 | 33 | 31
units | 6.06 [3.68 to 8.44] | 7.90 [4.95 to 10.85] | 8.56 [5.75 to 11.37]

3. Secondary Outcome: Number of Patients With Physicians Who Were Satisfied or Very Satisfied With Ease of Medication Administration
Description: This outcome is designed to examine MD satisfaction with ease of administration of intranasal medication - physicians who expressed that they were satisfied or very satisfied with ease of medication administration will be counted.
Time Frame: 60 minutes
Measure: Number; unit: participants
Arm/Group | 200 mcL VOA | 500 mcL VOA | 1000 mcL VOA
Number analyzed (Participants) | 32 | 33 | 31
participants | 13 | 30 | 30

ADVERSE EVENTS:
Time Frame: From time of administration of intranasal midazolam until emergency department discharge, an average of 1 hour.
Arm/Group | 200 mcL VOA | 500 mcL VOA | 1000 mcL VOA
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 4/33 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200 mcL VOA (N=32) | 500 mcL VOA (N=33) | 1000 mcL VOA (N=31)
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 — Vomiting after administration of intranasal midazolam
Inadequate sedation (Surgical and medical procedures) | 0 | 2 | 0 — Did not achieve sedation adequate for completion of laceration repair

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No